CLINICAL TRIAL: NCT07161596
Title: Oral Health Status and Oral Health Related Quality of Life of a Group of Hemophilic Egyptian Children Before and After an Oral Health Educational Program: A Before and After Study
Brief Title: Oral Health Status and Oral Health Related Quality of Life in a Group pf Egyptian Hemophilic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Hatem Abdelmoniem Ibrahim Atteya, Masters Student, Cairo University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: oral healthstatus & hemophilia
Record Dates: First submitted 2025-06-18; First posted 2025-09-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia
Keywords: oral hygiene index simplified; oral health related quality of life; oral health status; def; DMF; Hemophilic children
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: oral health educational program is used to measure the oral health status before and after
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemophilic children: oral health educational program as intervention (Experimental): An oral health educational program delivered to hemophilic Egyptian children as the main intervention guided by the oral and dental care instructions recommended by the American Academy of Pediatric Dentistry (AAPD) and the World Federation of Hemophilia (WFH), and the oral care program by the Egyptian society of hemophilia
  Interventions: Behavioral: oral health educational program
- hemophilic children: no oral health educational program (no intervention) (No Intervention): for ethical considerations; no intervention group will be given the oral health educational program after the follow up oral health status indices are measured

INTERVENTIONS:
Behavioral: oral health educational program — oral health educational program to the hemophilic children guided by the oral and dental care instructions provided by the AAPD and World federation of hemophilia oral care instructions
  Arms: hemophilic children: oral health educational program as intervention

SUMMARY:
aim of the study:

1. to assess, investigate, and compare the oral health status and oral health related quality of life of a group of hemophilic Egyptian children before and after an oral health educational program
2. evaluate the effectiveness of oral health educational programs on the oral health status of the Egyptian hemophilic children

benefits to patients: oral health awareness and change in the oral care levels with methods that match their health needs benefits to clinician: better understanding of the oral conditions associated with hemophilic patients, and their effects on oral health benefits to community: improvement of children's oral health, oral health awareness, promoting the importance of regular dental check ups for children with hemophilia

DETAILED DESCRIPTION:
In a non randomized clinical trial, Egyptian hemophilic children will be submitted to this trial to assess and measure their oral health status and oral health related quality of life prior to an oral health educational program. two groups will be formulated; the hemophilic group that will take the oral health educational program and the control group (other group) wont be taking the oral health educational program, then control will be given the oral health educational program after the follow up period for a better oral health in the hemophilic community. the oral health status will be recorded using two indices; DMF and def Caries indices and the oral hygiene index simplified (OHI-S) at baseline and at 8 months follow up period. bimonthly visits will be scheduled to check on the hemophilic children oral health and following up on given oral hygiene instructions. the oral health educational program is a tailored program guided by the American academy of pediatric dentistry, the oral considerations in the world federation of hemophilia , and oral care program of the Egyptian society of hemophilia in Egypt. diet counselling will be given. after the 8 months following the oral health educational program, oral health status and oral health related quality of life will be measured in both group and the results will be recorded. Aim of the study is a better oral health care and better understanding on how to apply oral hygiene measures correctly in hemophilic children.

ELIGIBILITY:
Inclusion Criteria:

* both sexes having hemophilia A,B or C
* no associated co morbid diseases
* mild, moderate and severe forms of hemophilia
* children whose parents agreed to participate in the study

Exclusion Criteria:

* patients with psychiatric disorders
* children whose parents refused to participate in the study
* patients using drugs( as cyclosporine, phenytoin) inducing periodontal problems

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
oral health status in Egyptian hemophilic children | baseline
  Oral Health Status
  1. Dental Caries in Permanent Teeth (Decayed, Missing, and Filled Teeth Index) The Decayed, Missing, and Filled Teeth index records the number of decayed, missing due to caries, and filled permanent teeth. A mean score is calculated for the study group.
     Mean DMFT score. Minimum value: 0 - Maximum value: 28. Higher scores indicate worse oral health status.
  2. Dental Caries in Primary Teeth (Decayed, Extracted, and Filled Teeth Index) The Decayed, Extracted, and Filled Teeth index records decayed, extracted due to caries, and filled primary teeth. A mean def score is reported for the study group.
     Minimum value: 0 - Maximum value: 20. Higher scores indicate worse oral health status.
  3. Oral Hygiene Status (Oral Hygiene Index-Simplified) The Oral Hygiene Index-Simplified combines debris and calculus scores to assess oral hygiene status Mean score.
  least value: 0 - Max:6 Lower score indicate better oral hygiene, and higher scores indicate worse oral hygiene.

SECONDARY OUTCOMES:
oral health related quality of life of a group of Egyptian hemophilic and non hemophilic children | baseline
  Oral Health-Related Quality of Life 4. CPQ11-14 Total Score The validated Arabic Child Perceptions Questionnaire (CPQ11-14) includes 36 items across four domains: oral symptoms, functional limitations, emotional well-being, and social well-being. The sum of all items provides a total score. Higher scores indicate greater negative impact.
  Unit of Measure: Mean CPQ11-14 total score (range 0-144) 5. CPQ11-14 Domain Scores Description: Sub scores are reported separately for oral symptoms, functional limitations, emotional well-being, and social well-being.
  Unit of Measure: Mean domain score (Oral symptoms: 0-24; Functional limitations: 0-36; Emotional well-being: 0-36; Social well-being: 0-48) 6. Global Rating of Oral Health Description: Children provide a self-assessment of oral health: excellent, very good, good, acceptable, or bad.
  Unit of Measure: Ordinal score (0 = excellent, 1 = very good, 2 = good, 3 = acceptable, 4 = bad) 7. Overall Well-Being Impact of Oral Health ordinal score

CONTACTS AND LOCATIONS:
Overall Officials: Nevine G Waly, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. No supporting documents will be made publicly available.

REFERENCES:
- See also: AL-KHAYAL, Z. and BROWN, A. (2006) 'Validity and reliability of the Arabic translation of the child oral-health-related quality of life questionnaire (CPQ11-14) in Saudi Arabia', Wiley Online Library. — https://pubmed.ncbi.nlm.nih.gov/17014538/.
- See also: Babu, N. S. Venkatesh, et al. (2016) 'Oral Health Status in Children with Haemophilia - a Comparative Study', The Journal of Haemophilia Practice, 3(2), pp. 43-47DOI: 10.17225/jhp00081. — https://sciendo.com/article/10.17225/jhp00081
- See also: Kabil, N., ElAlfy, M. S., and Metwalli, N. (2007) 'Evaluation of the oral health situation of a group of Egyptian haemophilic children and their re-evaluation following an oral hygiene and diet education programme', Haemophilia: The Official Journal of t — https://pubmed.ncbi.nlm.nih.gov/17498078/
- See also: Li, Y., et al. (2023) 'Oral health status and oral habits of children and adolescents with hemophilia: A report from the Children's Hemophilia Comprehensive Care Center of China', European Journal of Pediatrics, 183(2), pp. 897-902. — https://pmc.ncbi.nlm.nih.gov/articles/PMC10912247/